CLINICAL TRIAL: NCT00388648
Title: Efficacy and Safety of a Very Low Protein Diet in Postponing Dialysis in Elderly: a Prospective Randomized Multicenter Controlled Study
Brief Title: Very Low Protein Diet or Dialysis in Uremic Elderly?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NBs2000
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Uremia; Elderly (Aged >70); Dialysis; Low Protein Diet; Survival
Keywords: Dialysis; Vegan Diet; Mortality; Morbidity; Treatment outcome
MeSH Terms: conditions — Uremia | interventions — Keto Acids

INTERVENTIONS:
Drug: mixture of amino and keto acids

SUMMARY:
There are no solid data on the real advantage of an early start of dialysis, as suggested by the DOQI guidelines. Uremic patients frequently have a poor nutritional status. However, we cannot distinguish between the detrimental effect on nutrition of too low a residual renal function or too long a period of low protein-diet, per se. However, it appears that a very-low-protein diet (VLPD) supplemented with essential amino acids and keto-analogs of amino acids, and with an adequate quantity of calories, can prevent hypoalbuminemia at the start of dialysis and can slow the progression of chronic renal failure.

EDTA and USRDS data suggest that most patients starting dialysis nowadays are elderly, who also have the highest incidence of morbidity and mortality. Moreover, hospitalization rate becomes higher after the start of dialysis compared to the pre-dialysis period.

Can an aminoacid-supplemented VLPD, prolonged beyond the GFR limits suggested by DOQI, offer elderly patients better survival and better quality of life than dialysis? The answer can only come from a prospective, randomized trial, in elderly patients, starting at the GFR values suggested by the NKF-DOQI for starting dialysis, comparing outcomes with a vegetarian VLPD supplemented with a mixture of keto-analogs of amino acids and essential amino acids, and with dialysis.

DETAILED DESCRIPTION:
An adequate dose of dialysis is needed, in order to improve patient outcome, in both peritoneal dialysis (PD) and extracorporeal dialysis (HD). The debate, however, has renewed interest in when to start dialysis. The NKF-DOQI group suggested using the amount of solute clearance for regular dialysis as a value for starting dialysis treatment, i.e. creatinine clearance 9-14 ml/min.

Elderly patients on dialysis have a low survival rate.In fact, according to the lombard Registry(a italian region), patients 70-75 years old survive 2.9/3.6 years (male/female) after the start of dialysis, those 75-80 years old 2.7/2.7 years, and those 80-85 years old 2.4/1.4 years. This low survival is largely due to the combined effects of aging and comorbidities, on which an early start of dialysis has no or very limited positive effects.

Moreover, the hemodialytic treatment might have more negative effects in the elderly: intermittent hemodynamic stress, continuous fluctuation of electrolytes, metabolites, acid-base equilibrium, and the bioincompatibility of the membrane. In PD patients, the negative effects are also related to episodes of peritonitis and to daily loss of protein and a higher frequency of malnutrition.

An early start of dialysis should improve survival and well-being, and reduce morbidity. But a rapid decline of residual renal function (RRF) is observed after the start of dialysis. Maintenance of RRF as long as possible is very important, because the kidneys do some things a dialysis membrane cannot do: tubular and endocrine function, larger clearances of middle molecules, some of them potentially toxic such as parathyroid hormone, granulocyte inhibitory protein, and substances inducing anorexia.

In a prospective study on CAPD patients, for every increase of 1 ml/min of GFR, the relative risk (RR) of death decreased 50%. In the CanUsa study, using the time-dependent Cox multivariate analysis, a 5% reduction in RR of death was observed for each 5L/week of residual renal GFR at baseline (7). These results suggest that, at least in elderly patients, the fast decline of GFR observed after the start of dialysis could be another cause of the low survival rate.

In our center, 42 elderly patients started a very-low-protein diet (VLPD: 0.3 g of protein/kg body weight), supplemented with a mixture of keto acids and amino acids when their creatinine clearance reached values usually considered as a parameter for starting dialysis. The survival of this group of patients was compared with that of 71 patients directly put onto dialysis with the same creatinine clearance at which we started the VLPD. Subsequently, 24 patients in the diet group started dialysis when their mean GFR was 3.9 ml/min, i.e. lower than the 7 ml/min usually considered adequate in PD patients and much lower than 9-14 ml/min suggested by the NKF-DOQI group.

In this retrospective, non-randomized study, survival was better in the patients treated with diet than patients with dialysis. This seems to bear out that RRF does more than a dialytic membrane and must be preserved as long as possible.

ELIGIBILITY:
Inclusion Criteria:

1. males or females >= 70 years of age
2. RRF 5-7 ml/min/1.73 m2
3. left ventricular ejection fraction >40%
4. signed informed written consent

Exclusion Criteria:

1. diabetes
2. severe cerebral disease
3. proteinuria >3 g/24 h
4. severe hepatic failure
5. active malignancy
6. COPD requiring supplementary oxygen
7. AIDS, or HIV-positive

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160
Dates: Start 2000-01; Study Completion 2005-07

PRIMARY OUTCOMES:
The primary hypotheses to be tested are whether, at least in the elderly:
the supplemented Very Low Protein Diet (VLPD) does not increase the risk of morbidity and mortality,
a prolonged period of VLPD can postpone the need for dialysis in elderly patients, and dialysis can start at a RRF lower than usually suggested.

SECONDARY OUTCOMES:
the VLPD does not induce malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni c Cancarini, Prof, Study Chair — University of Brescia (Italy)
Locations (1):
- Dept of Nephrology, Brescia, Brescia, Italy

REFERENCES:
- [Result] Maiorca R, Brunori G, Viola BF, Zubani R, Cancarini G, Parrinello G, De Carli A. Diet or dialysis in the elderly? The DODE study: a prospective randomized multicenter trial. J Nephrol. 2000 Jul-Aug;13(4):267-70. PMID 10946805
- [Derived] Brunori G, Viola BF, Parrinello G, De Biase V, Como G, Franco V, Garibotto G, Zubani R, Cancarini GC. Efficacy and safety of a very-low-protein diet when postponing dialysis in the elderly: a prospective randomized multicenter controlled study. Am J Kidney Dis. 2007 May;49(5):569-80. doi: 10.1053/j.ajkd.2007.02.278. PMID 17472838